CLINICAL TRIAL: NCT03699943
Title: Feasibility Study of Intra-cavernosal Administration of Non-Expanded Autologous Bone Marrow Concentrate in Treatment of Erectile Dysfunction.
Brief Title: Autologous Bone Marrow Concentrate in Treatment of Erectile Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creative Medical Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 21511-01
Record Dates: First submitted 2015-12-12; First posted 2018-10-09 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Caverstem 1.0 - Low dose - 30 cc - 20 patients Caverstem 1.0 - High dose - 60 cc - 20 patients Caverstem 2.0 - 20 cc - 100 patients
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CaverStem 1.0 - Low (Active Comparator): Intra-cavernosal injection of autologous bone marrow concentrate for the treatment of Erectile Dysfunction. low dose 30 cc
  Interventions: Procedure: CaverStem
- CaverStem 1.0 - High (Active Comparator): Intra-cavernosal injection of autologous bone marrow concentrate for the treatment of Erectile Dysfunction. high dose 60 cc
  Interventions: Procedure: CaverStem
- Caverstem 2.0 - Clinical Registry (Active Comparator): Intra-cavernosal injection of autologous bone marrow concentrate for the treatment of Erectile Dysfunction. 20 cc
  Interventions: Procedure: CaverStem

INTERVENTIONS:
Procedure: CaverStem

SUMMARY:
This study assessed the safety and efficacy of autologous bone marrow concentrate and injected intra-cavernously into patients with erectile dysfunction (ED). Specifically, this study will evaluate ED treatment >18 year old men, a demographic where the etiology of ED is attributable primarily to the loss of corporal smooth muscle in the penis. Study endpoints will evaluate the safety and efficacy of intracavernosal bone marrow concentrate administration for treating ED patients.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is characterized by abnormalities of the vascular system; most commonly, venous leakage (or veno-occlusive dysfunction) resulting from loss of integrity of the surrounding corporal smooth muscle. In the penile vascular system, the corporal smooth muscle is responsible for trapping the blood delivered to the corpora cavernosa via the arterial system.

Bone marrow is enriched for cells with regenerative potential, including mesenchymal stem cells, which accelerate healing of damaged tissue. The possibility of using bone marrow cells in the treatment of ED is enticing since stem/progenitor cell populations are known to secrete various growth factors, possess anti-inflammatory activities, and can differentiate into cells of the penile architecture.

This study will evaluate safety and efficacy of autologous bone marrow concentrate generated by a closed system device and injected intra-cavernously in 40 patients aged > 18 years of age diagnosed with erectile dysfunction with low dose 30 cc (20 patients) or high dose 60 cc (20 patients). Safety and efficacy will be evaluated at baseline (prior to treatment) and at 1,3,6 and 12-month follow up visits. The study will determine whether injection of bone marrow cells intra-cavernously is a clinically feasible, safe and reproducible approach for treating erectile dysfunction. A clinical registry will also be enrolling treating the same patient population (100 patients (20 cc)).

ELIGIBILITY:
Inclusion Criteria:

1. Chronic organic ED duration at least 0.5 years
2. Diagnosis of ED based on Doppler Ultrasound and/or dynamic infusion cavernosonometry.
3. Baseline International Index of Erectile Function (IIEF-5) score of < 21
4. Oral medications and intracavernous pharmacological approaches have been deemed ineffective, contraindicated or cannot be tolerated.
5. Concurrently undergoing treatment with testosterone.
6. Willing to forego any other treatments for ED over the course of the study.

Exclusion Criteria:

1. Subjects using any medications/drugs with known effects on erectile function within 4 weeks of the study period, including certain antidepressants, antihistamines, diuretics, and beta-blockers.
2. Subjects using herbal remedies for addressing erectile dysfunction within one month of study initiation.
3. Subjects with penile prosthesis or other urinary prosthesis.
4. Subjects with penile anatomical deformities (e.g. Peyronie's disease) or history of priapism.
5. Previous penile surgeries for erectile dysfunction, premature ejaculation or penile enlargement.
6. Diagnosis of psychogenic ED as determined by nocturnal tumenscence testing.
7. Presenting with uncontrolled or severe disease, including cardiovascular disease, diabetes, liver disease.
8. Uncontrolled hypertension or hypotension (systolic blood pressure > 170 or < 90 mm Hg, and diastolic blood pressure > 100 or < 50 mm Hg)
9. Suffered a cardiovascular event within 6 months prior to study initiation.
10. Current or previous malignancy other than non-melanoma skin cancer (successfully treated or treatable by curative excision or other local curative therapy).
11. Diagnosis of a systemic autoimmune disorder.
12. Receiving immunosuppressant medications.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Improvement in erectile function as measured by total score in the International Index of Erectile Function | 6 months
  IIEF-5 scale
Rate of Adverse Events | 6 months
  bruising, infection, pain

SECONDARY OUTCOMES:
Change in Doppler Measurements | 6 months
  ml/s

CONTACTS AND LOCATIONS:
Overall Officials: Alex Gershman, Study Chair — UCLA/Cedar; Jacob Rajfer, Study Director — University of California, Los Angeles
Locations (1):
- Harbor - UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared among other investigators through secure clinical registry.
Supporting Information: SAP, ICF, CSR
Time Frame: 1 year

REFERENCES:
- [Derived] Bieri M, Said E, Antonini G, Dickerson D, Tuma J, Bartlett CE, Patel AN, Gershman A. Phase I and registry study of autologous bone marrow concentrate evaluated in PDE5 inhibitor refractory erectile dysfunction. J Transl Med. 2020 Jan 14;18(1):24. doi: 10.1186/s12967-019-02195-w. PMID 31937310